CLINICAL TRIAL: NCT01296412
Title: A Phase III, Multicenter, Randomized, Open-label Clinical Trial Comparing the Efficacy and Safety of a Sitagliptin-Based Treatment Paradigm to a Liraglutide-Based Treatment Paradigm in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin Monotherapy
Brief Title: Comparison of Two Treatment Regimens (Sitagliptin Versus Liraglutide) on Participants Who Failed to Achieve Good Glucose Control on Metformin Alone (MK-0431-403)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0431-403
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Results first posted 2013-03-15 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Liraglutide; glimepiride; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin +/- glimepiride (Experimental): Sitagliptin 100 mg tablet orally once daily for 26 weeks. Participants continued their stable dose of metformin >=1500 mg orally daily. Participants may have received glimepiride orally for glycemic control.
  Interventions: Drug: sitagliptin; Drug: glimepiride; Drug: metformin
- Liraglutide (Active Comparator): Liraglutide subcutaneous injection once daily for 26 weeks (starting dose 0.6 mg daily up-titrated to 1.2 mg daily on Day 8). Participants continued their stable dose of metformin >=1500 mg orally daily. Participants may have had their liraglutide dose uptitrated to 1.8 mg daily for glycemic control.
  Interventions: Drug: liraglutide; Drug: metformin

INTERVENTIONS:
Drug: sitagliptin — 100 mg tablet, orally, once daily.
  Other Names: MK-0431, Januvia®, Tesavel®, Xelevia®, Ristaben®
  Arms: Sitagliptin +/- glimepiride
Drug: liraglutide — 0.6 mg by subcutaneous (pen) injection, once daily, on Days 1-7; up-titrated on Day 8 to 1.2 mg daily. At Week 12, dose may be increased to 1.8 mg once daily for participants who did not meet protocol-specified glycemic goals.
  Other Names: Victoza®
  Arms: Liraglutide
Drug: glimepiride — starting dose of 1 mg tablet (up-titrated as needed), once daily, as needed, after Week 12.
  Other Names: Amaryl®
  Arms: Sitagliptin +/- glimepiride
Drug: metformin — metformin tablets at a dose of ≥1500 mg per day
  Other Names: Fortamet®, Glucophage®, Glucophage® XR, Glumetza®, Riomet®, Metgluco®, Glycoran®

SUMMARY:
This study is being done to compare the effectiveness and safety of two treatment paradigms (oral sitagliptin with or without glimepiride versus liraglutide with or without increased dosing) for the treatment of participants with Type 2 Diabetes that is not adequately controlled with metformin alone. The primary hypothesis postulated that the mean change from baseline in hemoglobin A1c (A1C) in participants treated with a sitagliptin-based treatment is non-inferior to that of participants treated with a liraglutide-based

treatment.

ELIGIBILITY:
Inclusion criteria

* Type 2 diabetes mellitus.
* On stable dose of metformin monotherapy at a dose of at least 1500 mg per day for at least 12 weeks and a hemoglobin A1C ≥7.0% and ≤11.0%.
* Capable of using a liraglutide pen device.

Exclusion criteria

* History of Type 1 Diabetes mellitus.
* Use of any oral antihyperglycemic agent (AHA) besides metformin, within the prior 12 weeks of screening.
* Cardiovascular disorders within the past 3 months including acute coronary syndrome or new or worsening symptoms of coronary heart disease, coronary artery intervention, stroke, or transient ischemic neurological disorder.
* Impaired liver function.
* Impaired kidney function.
* History of malignancy or clinically important hematological disorder that requires disease-specific treatment (chemotherapy, radiation therapy, surgery) or, in the opinion of the investigator, is likely to recur during the duration of the study.
* History of leukemia, lymphoma, aplastic anemia, myeloproliferative or myelodysplastic diseases, thrombocytopenia, or malignant melanoma, regardless of the time since treatment.
* Pregnancy or breastfeeding, or intention to become pregnant or donate eggs within the projected duration of the study.
* Participation in another study with an investigational drug or device within 12 weeks prior to screening.
* History of hypersensitivity or any contraindication to sitagliptin, liraglutide, glimepiride, or metformin based upon the labels of the country of the investigational site.
* Participation in a weight loss program and not yet in maintenance phase, or starting of a weight loss medication (such as orlistat or phentermine) within the prior 8 weeks.
* Surgery within the prior 4 weeks or major surgery planned during the study.
* Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN 2).
* User of recreational or illicit drugs or recent history (within the last year) of drug abuse or increased alcohol consumption.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 653 (Actual)
Dates: Start 2011-03-11 (Actual); Primary Completion 2012-02-29 (Actual); Study Completion 2012-02-29 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Charbonnel B, Steinberg H, Eymard E, Xu L, Thakkar P, Prabhu V, Davies MJ, Engel SS. Efficacy and safety over 26 weeks of an oral treatment strategy including sitagliptin compared with an injectable treatment strategy with liraglutide in patients with type 2 diabetes mellitus inadequately controlled on metformin: a randomised clinical trial. Diabetologia. 2013 Jul;56(7):1503-11. doi: 10.1007/s00125-013-2905-1. Epub 2013 Apr 19. PMID 23604551

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitagliptin +/- Glimepiride: Sitagliptin 100 mg tablet once daily for 26 weeks. Participants continued their stable dose of metformin >=1500 mg orally daily. Participants may have received glimepiride for glycemic control.
Period: Overall Study
Arm/Group | Sitagliptin +/- Glimepiride | Liraglutide
Started | 326 | 327
Completed | 275 | 257
Not Completed | 51 | 70
Not completed — Adverse Event | 8 | 29
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 10 | 7
Not completed — Non-compliance with study drug | 1 | 2
Not completed — Other reason not specified | 20 | 15
Not completed — Physician Decision | 1 | 3
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal by Subject | 10 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin +/- Glimepiride | Liraglutide | Total
Number analyzed (Participants) | 326 | 327 | 653
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (10.0) | 57.6 (10.8) | 57.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 147 | 295
  Male | 178 | 180 | 358
Hemoglobin A1c (A1C) [Mean (Standard Deviation); unit: Percent] — A1C baseline values are presented for participants with data: Sitagliptin + metformin, n=325; liraglutide + metformin, n= 325; total population, n=650
  Percent | 8.2 (1.1) | 8.1 (0.9) | 8.2 (1.0)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] — FPG baseline values are presented for participants with data: Sitagliptin + metformin, n=325; liraglutide + metformin, n= 325; total population, n=650
  mg/dL | 174.1 (43.7) | 172.9 (40.8) | 173.5 (42.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (A1C)
Description: A1C is measured as percent. Thus, this change from baseline reflects the Week 26 A1C percent minus the Week 0 A1C percent.
Time Frame: Baseline and Week 26
Population: Per-protocol population defined as participants who had a measurement at baseline and a measurement after at least 24 weeks (i.e., 168 days) of treatment, and did not have any major protocol violations.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Sitagliptin +/- Glimepiride | Liraglutide
Number analyzed (Participants) | 269 | 253
percent | -1.32 (1.06) [-1.42 to -1.23] | -1.42 (1.04) [-1.51 to -1.32]
Statistical Analysis 1: Comparison: Sitagliptin +/- Glimepiride vs Liraglutide; Test type: Non-Inferiority or Equivalence — The sitagliptin-based treatment paradigm was to be declared non-inferior to the liraglutide-based treatment paradigm in lowering A1C at Week 26 if the upper bound of 95% confidence intervals of between group difference was less than the non-inferiority margin of 0.4%; ANCOVA; The ANCOVA model included a term for treatment paradigm and a covariate for baseline value; Difference in least squares mean = 0.09, 95% CI 2-sided [-0.05 to 0.23]

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Change from baseline at Week 26 is defined as Week 26 minus Week 0.
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin +/- Glimepiride | Liraglutide
Number analyzed (Participants) | 269 | 252
mg/dL | -33.7 (46.2) [-37.5 to -29.9] | -39.6 (40.3) [-43.6 to -35.7]
Statistical Analysis 1: Comparison: Sitagliptin +/- Glimepiride vs Liraglutide; Test type: Superiority or Other; ANCOVA; The ANCOVA model included a term for treatment paradigm and a covariate for baseline value; Difference in least squares mean = 5.9, 95% CI 2-sided [0.5 to 11.4]

3. Secondary Outcome: Percentage of Participants Reaching A1C Goal of <7.0%
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Sitagliptin +/- Glimepiride | Liraglutide
Number analyzed (Participants) | 269 | 253
percentage of participants | 62.8 | 72.3
Statistical Analysis 1: Comparison: Sitagliptin +/- Glimepiride vs Liraglutide; Test type: Superiority or Other; Miettinen & Nurminen; Difference in percent = -9.5, 95% CI 2-sided [-17.4 to -1.5]

4. Secondary Outcome: Percentage of Participants Reaching A1C Goal of <6.5%
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Sitagliptin +/- Glimepiride | Liraglutide
Number analyzed (Participants) | 269 | 253
percentage of participants | 33.8 | 38.3
Statistical Analysis 1: Comparison: Sitagliptin +/- Glimepiride vs Liraglutide; Test type: Superiority or Other; Miettinen & Nurminen; Difference in percent = -4.5, 95% CI 2-sided [-12.7 to 3.7]

ADVERSE EVENTS:
Description: Safety analyses were performed on the all participants as treated population (defined as participants who received at least 1 dose of study therapy). Participants were included in the reporting group corresponding to the actual study treatment received. Three participants randomized to therapy did not receive any study therapy.
Arm/Group | Sitagliptin +/- Glimepiride | Liraglutide
Serious Adverse Events (participants affected / at risk) | 17/326 | 12/324
Other Adverse Events (participants affected / at risk) | 58/326 | 97/324
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin +/- Glimepiride (N=326) | Liraglutide (N=324)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Accidental death (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subcutaneous hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (2)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blue toe syndrome (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin +/- Glimepiride (N=326) | Liraglutide (N=324)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 35 (42)
Nausea (Gastrointestinal disorders) | 10 (13) | 63 (73)
Vomiting (Gastrointestinal disorders) | 6 (10) | 21 (25)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 21 (21)
Hypoglycaemia (Metabolism and nutrition disorders) | 41 (89) | 15 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.